CLINICAL TRIAL: NCT02596594
Title: Intraumbilical Amino Acids and Glucose Supplementation Via Subcutaneously Implanted Port System by Severe IUGR Human Fetuses
Brief Title: Intraumbilical Amino Acids and Glucose Supplementation Via Port by Severe IUGR in Human Fetuses
Acronym: port-IUGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Michael Tchirikov MD, PhD, MD PhD, Martin-Luther-Universität Halle-Wittenberg
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 110; 3/15-08-2012
Record Dates: First submitted 2015-10-12; First posted 2015-11-04 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Intrauterine Growth Restriction
Keywords: IUGR; severe IUGR; brain sparing; fetal nutrition; Prolongation; pregnancy; neonatal outcome
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Intraumbilical amino acid and glucose suplementation of human fetuses with a severe IUGR via a subcutaneously implanted port system
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Port intervention (Experimental): The subcutaneous intraumbilical port-system will be implanted in IUGR patients with the cerebroplacental ratio less than 1 (cerebroplacental ratio= PI in the middle cerebral artery / PI umbilical artery) between 24/0 and 30/0 weeks of gestation.
  The fetuses will receive AAs and glucose supplementation via a subcutaneously implanted intraumbilical perinatal port system till the delivery. Control by doppler and cardiotocogram
  Interventions: Device: fetal nutrition port system
- control (No Intervention): IUGR patients with the cerebroplacental ratio less than 1 (CPR= PI middle cerebral artery / PI umbilical artery) between 24/0 and 30/0 weeks of gestation.
  Control by doppler and cardiotocogram

INTERVENTIONS:
Device: fetal nutrition port system — Under local anesthesia a subcutaneous pouch for the port capsule was prepared using a pair of scissors. The umbilical vein was punctured with a 18 gauge needle under ultrasound control and the catheter was inserted into the umbilical vein. Note the amniotic cavity remained intact. A 25 gauge port needle was used to enter the port system. The treatment course included daily infusions of AA solution (Fresenius Kabi, Bad Homburg, Germany) with a 10% glucose solution. The investigators limited the volume of the intraumbilical infusion to 10% of the estimated feto-placental blood volume per day. On average, the AA/glucose-infusion was below 50 ml/kg.
  Arms: Port intervention

SUMMARY:
Placental insufficiency is responsible for fetal loss in about 40% of all stillbirths and long term neurological deficits. The mean interval from diagnosis of brain sparing of severe IUGR fetuses to delivery has been recently identified by only seven days (Flood K et al, Am J Obstetrics and Gynecology 2014).

The critical placental player in the active amino acids (AA) transport from the mother to the fetus is the trophoblast, which is irreversibly changed in severe IUGR fetuses caused by placental insufficiency. Thus, a logical partial solution of IUGR could be the direct supply of AAs and glucose to the fetus, in order to improve the fetal growth, normalize the fetal programming and to prolong the pregnancy.

The aim of this prospective pilot study is to further test the efficacy of the administration of AAs and glucose supplementation with hyperbaric oxygenation (HBO), via a subcutaneously implanted intraumbilical perinatal port system, as a treatment option for severe IUGR human fetuses with brain sparing.

DETAILED DESCRIPTION:
Placental insufficiency is the main source of the development of intrauterine growth restriction (IUGR) caused by one of a variety of factors including chronic placental infections, many maternal diseases, abnormal genome and intravascular trophoblast invasion impairment. Placental insufficiency is responsible for fetal loss in about 40% of all stillbirths and long term neurological deficits. The reduction of blood flow resistance of cerebral arteries in severe IUGR conditions with reduced pulsatility index (PI) in the medial cerebral artery predicts the 11 fold increased risk of intraventricular hemorrhage, periventricular leukomalacia, hypoxic ischemic encephalopathy, necrotizing enterocolitis, bronchopulmonary dysplasia, sepsis, and death. The mean interval from diagnosis of brain sparing of severe IUGR fetuses to delivery has been recently identified by only seven days (ranging 2-15 days).

The amino acids (AA) concentration of fetal plasma is many times higher than in mother because of active transplacental transport of AA and additional AA synthesis in the placenta.

The critical placental player in the active AA transport from the mother to the fetus is the trophoblast, which is irreversibly changed in severe IUGR fetuses caused by placental insufficiency. Thus, a logical partial solution of IUGR could be the direct supply of AAs and glucose to the fetus, in order to improve the fetal growth, normalize the IUGR changed fetal programming and to prolong the pregnancy. Additional oxygen supply of fetal tissues could also be important in improving the uptake of injected nutritional supplements and may avoid the development of lactate acidosis in IUGR fetuses.

The aim of this prospective pilot study was to further test the efficacy of the administration of AAs and glucose supplementation with hyperbaric oxygenation (HBO), via a subcutaneously implanted intraumbilical perinatal port system, as a treatment option for severe IUGR human fetuses with brain sparing.

Study design - IUGR was defined in this study as an estimated fetal weight of < 5%, combined with increased resistance in both uterine arteries with pulsatility index (PI) > 95%. Fetuses with morphological and/or chromosomal abnormalities were not included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of severe intrauterine growth restricted fetuses with the cerebroplacental ratio less than 1 (CPR= PI middle cerebral artery / PI umbilical artery)
2. gestational age between 24/0 and 30/0 weeks
3. single pregnancy
4. anterior or lateral location of the placenta

Exclusion Criteria:

1. multiple pregnancy
2. fetal genetic anomalities,
3. fetal morphologic anomalities
4. BMI > 35
5. placenta praevia
6. vaginal bleeding
7. uterine contractions
8. vasa praevia
9. posterior location of the placenta
10. severe maternal morbidities
11. Infections
12. preliminary rupture of the membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The mean interval from diagnosis of brain sparing of severe IUGR fetuses to delivery | through study completion, up to 2 years
  The mean interval from diagnosis of brain sparing of severe IUGR fetuses to delivery will be documented (days). The timing of delivery by caesarean section will be decided by the lead clinician managing each case based on doppler and cardiotocogram clinical evaluations.

SECONDARY OUTCOMES:
neonatal weight | through study completion, up to 2 years
  the neonates' weight will be estimated after the delivery
fetal weight gain | through study completion, up to 2 years
  the difference (g) between estimated by ultrasound fetal weight and neonatal weight at delivery
blood gas analysis in the umbilical artery | through study completion, up to 2 years
  the blood gas analysis in the umbilical artery will be performed after the delivery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tchirikov, MD, PhD, Principal Investigator — Martin-Luther University Halle-Wittenberg

REFERENCES:
- [Background] Tchirikov M, Kharkevich O, Steetskamp J, Beluga M, Strohner M. Treatment of growth-restricted human fetuses with amino acids and glucose supplementation through a chronic fetal intravascular perinatal port system. Eur Surg Res. 2010;45(1):45-9. doi: 10.1159/000318859. Epub 2010 Aug 20. PMID 20733317